CLINICAL TRIAL: NCT06094179
Title: A Study Evaluated the Safety and Efficacy of BAT6026 in Patients With Moderate to Severe Atopic Dermatitis Phase I/II Clinical Study
Brief Title: Evaluate the Safety, Tolerability of BAT6026
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BAT-6026-003-CR
Record Dates: First submitted 2023-10-08; First posted 2023-10-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a Phase IB/IIA clinical study of BAT6026 in patients with AD. The subjects were adults with moderate to severe atopic dermatitis (AD) whose disease was not adequately controlled by prior topical medications or for which topical medications were not appropriate. The first phase was the phase IB study, which was double-blind controlled by placebo in the group and consisted of 3 dose groups. After completing the dose escalation study, the phase IIA study was entered. The Phase IIA study was a randomized, double-blind, controlled, multicentering clinical trial with different dose groups and placebo groups. The primary endpoint was to explore the efficacy and safety of BAT6026 in patients with eczema area and severity index (EASI) of at least 75% lower than the baseline at week 16 after 4 treatment cycles. To provide the optimal dose for the phase III regimen.
Who Masked: Participant, Investigator
Masking Description: Phase IB and Phase IIA of this study were double-blind trials. Neither the subject nor the investigator nor the sponsor's project team members were aware of the subject's treatment assignment. Supply of the investigational drug and placebo by the sponsor or designated unit. To reduce the likelihood of subjects being exposed to unnecessary risks while providing the necessary information for dosing escalation, discontinuation and selection, a Safety Management Committee (SMC) will be established to review the subject safety data as necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A1 300mg (Experimental): Trial drug: Placebo 9:3 randomized double-blind admission. The last patient in each group was given the drug for 1 week, and the existing safety data was reviewed blind by SMC, and the next group was entered into the study after reaching the increasing standard
  Interventions: Drug: Monoclonal antibody BAT6026; Drug: sodium chloride injection
- B1 600mg (Experimental): Trial drug: Placebo 9:3 randomized double-blind admission. The last patient in each group was given the drug for 1 week, and the existing safety data was reviewed blind by SMC, and the next group was entered into the study after reaching the increasing standard
  Interventions: Drug: Monoclonal antibody BAT6026; Drug: sodium chloride injection
- C1 600mg (Experimental): Trial drug: Placebo 9:3 randomized double-blind admission. The last patient in each group was given the drug for 1 week, and the existing safety data was reviewed blind by SMC, and the next group was entered into the study after reaching the increasing standard
  Interventions: Drug: Monoclonal antibody BAT6026; Drug: sodium chloride injection

INTERVENTIONS:
Drug: Monoclonal antibody BAT6026 — 300mg Q4W group, 600mg Q4W group (at week 0,4,8,12) and 600mg Q2W group (at week 0,2,4,6,8,10,12,14)
  Other Names: BAT6026
Drug: sodium chloride injection — 300mg Q4W group, 600mg Q4W group (at week 0,4,8,12) and 600mg Q2W group (at week 0,2,4,6,8,10,12,14)

SUMMARY:
This is a Phase IB/IIA clinical study of BAT6026 in patients with AD. The subjects were adults with moderate to severe atopic dermatitis (AD) whose disease was not adequately controlled by prior topical medications or for which topical medications were not appropriate. The first phase was the phase IB study, which was double-blind controlled by placebo in the group and consisted of 3 dose groups. After completing the dose escalation study, the phase IIA study was entered. The Phase IIA study was a randomized, double-blind, controlled, multicentering clinical trial with different dose groups and placebo groups. The primary endpoint was to explore the efficacy and safety of BAT6026 in patients with eczema area and severity index (EASI) of at least 75% lower than the baseline at week 16 after 4 treatment cycles. To provide the optimal dose for the phase III regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign written informed consent and comply with the requirements of the research protocol;
2. age 18-75 years old, male and female;
3. According to the Hanifin-Rajka criteria, the patient was diagnosed with AD and had a history of at least 1 year;
4. EASI score ≥16 during screening visit and baseline visit;
5. IGA score ≥3 at screening and baseline (moderate);
6. BSA involvement at screening and baseline was ≥10%;
7. Received glucocorticoids, phosphodiesterase inhibitors, or calcineurin inhibition in the 6 months prior to screening Drug, or phototherapy for AD and other local treatment options, and according to the judgment of the investigator, the local treatment response is insufficient (follow the doctor Local treatment is prescribed for at least 4 weeks or to the maximum recommended course of treatment in the product's prescribing information, whichever is shorter, which has not been achieved Is in remission or in a state of low disease activity (IGA 0 to 2), has no response or intolerance, or has a medical contraindication to the treatment, and is not suitable for the use of this local treatment;
8. Steady-dose topical emollients (subjects must use investigator-recommended or investigator-approved base emollients that do not contain AD-affecting additives, such as hyaluronic acid, urea, ceramide, or filagmin) have been applied for at least 7 consecutive days prior to baseline visit and continued use during the study period; If the patient is screened before the visit has been started These moisturizers can then be used in steady doses;
9. For women of childbearing age, it should not be during pregnancy or lactation; And all the subjects and their partners were in treatment

Exclusion Criteria:

1. Other inflammatory diseases that may confuse the diagnosis of AD or interfere with the evaluation of efficacy (e.g. Psoriasis, systemic erythematosus) Sore, scleroderma, mixed connective tissue disease, overlapping syndrome, etc.);
2. any of the following laboratory test abnormalities existed before the first drug use (individual indicators during the screening period do not meet, rescreening qualified can still be accepted

   In) :
   1. Hemoglobin <100 g/L;
   2. White blood cell count (WBC) <3.5×109/L;
   3. Neutrophil count <1.5×109/L;
   4. Platelet count <100×109/L;
   5. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2× upper limit of normal (ULN);
   6. Total bilirubin >1.5×ULN;
   7. Creatinine >1.2×ULN.
   8. abnormalities in other laboratory tests that, as determined by the investigator, may affect the completion or evaluation of the test;
3. Have a history of alcohol or drug abuse, alcoholism or drug dependence within 1 year before screening; Poor compliance as assessed by the investigator (approved Inquire);
4. Previous history of allergy to biological products or allergic to BAT6026 or any of its excipients;
5. within 6 months before the first drug, did not receive standard treatment (SOC) or SOC failed to infected parasites;
6. Systematic administration of antibiotics, antiviral drugs, antiparasitic drugs, antigenics or antigenics is required within 4 weeks before the first medication Antimicrobials are used to treat a variety of systemic infections, and the medical history assessed by the investigator or sponsor may interfere with subjects in this trial Safety, and efficacy evaluators;
7. have severe liver, kidney, hematology, gastrointestinal, endocrine, lung, heart, central nervous system or sperm God disease;
8. Patients with unstable or uncontrollable hypertension/diabetes need to be excluded, such as those who can be controlled and stabilized by drug treatment The researcher judged that it could continue to be included;
9. Superficial skin infection exists within 2 weeks before the first medication;
10. Received live vaccine within 4 weeks before the first dose, except inactivated vaccine;
11. Participated in any clinical trials 4 weeks before the first medication;
12. Received systemic glucocorticoids and other immunizations within 4 weeks or 5 half-lives (whichever is older) prior to the first dose Epidemic inhibitor therapy (e.g., cyclosporine, mycophenolate, interferon gamma, azathioprine, methotrexate, JAK enzyme suppression) Preparations), biological agents;
13. Receive any of the following topical drugs for AD within 1 week before the first dose:

    Glucocorticoids (TCS); Calcineurin inhibitors or other immunosuppressants; JAK inhibitor; Antipruritic agents such as clomitone; Compound preparations containing corticosteroids or calcineurin inhibitors or other immunosuppressants; Prescription emollients that affect AD; Chinese herbal medicine, proprietary Chinese medicine and ethnic medicine for AD;
14. Received natalizumab or other regulatory B or T cells within 12 months prior to the first dose Drug therapy, such as rituximab, alemtuzumab, abacil (abatacept), etc.
15. Received whole-body phototherapy (narrow-spectrum ultraviolet B [NB-UVB], ultraviolet B [UVB], Ultraviolet A [UVA], psoralen combined with ultraviolet A [PUVA])
16. Patients who had received major surgery within 4 weeks prior to the first dose or planned to undergo major surgery during the study period, or were unable to undergo surgery before randomization Complete recovery during operation;
17. patients with a history of malignant tumors (completely cured cervical carcinoma in situ, non-metastatic skin squamous cell carcinoma, skin Other than basal cell carcinoma), or lymphoproliferative diseases;
18. Patients who have received organ transplantation within 3 months before screening (corneal transplantation >3 months before the first administration of the experimental drug) External);
19. Pregnant or lactating women, or women who wish to become pregnant;
20. there are infected with the following diseases: active hepatitis B virus infection [Hepatitis B surface antigen (HBsAg) positive, and B Hepatovirus deoxyribonucleic acid (HBV-DNA) test >200 IU/ml or 103 copies /ml; Infected with hepatitis C virus [Positive results of HCV antibody and viral ribonucleic acid (HCV-RNA) detection]; Treponema pallidum antibody positive and RPR Positive or other confirmed tests;
21. Active tuberculosis includes, but is not limited to, tuberculosis (TB) in patients who have been treated with standardized anti-TB therapy and have been confirmed cured by researchers Included) and patients with latent tuberculosis (positive for Tspot or Quantiferon); History of immunodeficiency, including human immunity A history of HIV infection or other immunodeficiency diseases;
22. Those who have participated in OX40 antibody research and used OX40 antibody before;
23. Other conditions deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
tolerance | The last patient in each group was dosed 1 week later
  Incidence of AE above 3 Arms associated with the test drug in each dose group
Vital signs | The last patient in each group was dosed 1 week later
  Number of participants with abnormal vital signs
ECG parameters | The last patient in each group was dosed 1 week later
  Number of participants with abnormal ECG readings
Laboratory tests | The last patient in each group was dosed 1 week later
  Number of participants with abnormal laboratory test results
AEs, adverse events | The last patient in each group was dosed 1 week later
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Jianzhong Zhang, Beijing, Beijing Municipality, China